CLINICAL TRIAL: NCT02074358
Title: A Study to Assess the Effects of 2 Prothrombin Complex Concentrates on the Pharmacodynamics of Apixaban in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CV185-156; 2013-000646-18 (EudraCT Number)
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Results first posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-07

CONDITIONS: Anticoagulation
MeSH Terms: interventions — apixaban; prothrombin complex concentrates; factor IX, factor VII, factor X, prothrombin drug combination; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A: Apixaban + Placebo (Saline solution) (Experimental): Apixaban 10 mg Tablet orally [Day 1-Day 3: twice daily (BID), Day 4: Single Dose (SD)] followed 3hr later by Saline solution (placebo) 0 IU/kg infusion for 30 min Intravenously
  Interventions: Drug: Apixaban; Drug: Placebo (Saline solution)
- Treatment B: Apixaban + Cofact (4-Factor PCC) (Experimental): Apixaban 10 mg Tablet orally [Day 1-Day 3: twice daily (BID), Day 4: Single Dose (SD)] followed 3hr later by a Cofact (4-Factor PCC) 50 IU/kg infusion for 30 min Intravenously
  Interventions: Drug: Apixaban; Drug: Cofact (4-Factor PCC)
- Treatment C: Apixaban + Beriplex P/N (4-Factor PCC) (Experimental): Apixaban 10 mg Tablet orally [Day 1-Day 3: twice daily (BID), Day 4: Single Dose (SD)] followed 3hr later by a Beriplex P/N (4-Factor PCC) 50 IU/kg infusion for 30 min Intravenously
  Interventions: Drug: Apixaban; Drug: Beriplex P/N (4-Factor PCC)

INTERVENTIONS:
Drug: Apixaban
  Other Names: BMS-562247
Drug: Cofact (4-Factor PCC)
  Arms: Treatment B: Apixaban + Cofact (4-Factor PCC)
Drug: Beriplex P/N (4-Factor PCC)
  Arms: Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Drug: Placebo (Saline solution)
  Arms: Treatment A: Apixaban + Placebo (Saline solution)

SUMMARY:
The purpose of this study is to assess the effect of two 4-Factor PCC formulations on Apixaban pharmacodynamics in healthy adult subjects.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy subjects
* Body Mass Index (BMI) of 18 to 30 kg/m2
* Ages 18 to 45 years, including
* Women of childbearing potential (WOCBP) on acceptable contraception and with negative pregnancy test and not breastfeeding

Exclusion Criteria:

* History or evidence of coagulopathy
* History or evidence of thrombosis such as deep vein thrombosis or other thromboembolic disease or having a first degree relative under 50 years of age with a history of thromboembolic disease
* Any significant acute or chronic medical illness or relevant trauma
* Any major surgery within 4 weeks of dosing (prior to dosing) or planned within 2 weeks after completion of the study
* History of heavy menstrual bleeding that has produced anemia within the past 1 year
* Current symptomatic or recent gastrointestinal disease or surgery that could impact the absorption of study drug
* History of smoking within 1 month prior to dosing
* Recent history (within 6 months of dosing) of pregnancy
* Use of hormonal contraceptives
* Exposure to any investigational drug or placebo within 4 weeks of study drug administration
* Use of any agent, including but not limited to Aspirin, Nonsteroidal anti-inflammatory drugs (NSAIDs), Anticoagulants, Fish oil capsules, Gingko, etc, that are known to increase the potential for bleeding, within 2 weeks prior to dosing
* History of any severe drug allergy including allergy to Heparin or history of Heparin-induced thrombocytopenia, hypersensitivity to PCCs or Factor Xa inhibitors, or history of allergy to human blood plasma derived products; history of any adverse drug reaction to Anticoagulants or Antiplatelet agents that resulted in excessive bleeding requiring medical intervention

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study initiated in February 2014 in healthy adult participants and completed in April 2014. Participants were admitted to a clinical facility on the evening prior to dosing and remained in the facility for at least 72 hours after the start of the IV infusion on Day 4.
Pre-assignment Details: 43 enrolled;15 treated. Reasons not treated: 5 withdrew consent; 19 no longer met study criteria; 4 stand-by participants not needed (cohort full). Crossover: 6 treatment sequences (3 periods) with an 11 day washout from study drug between each treatment period; 3 participants in each sequence: ABC, ACB, CAB and 2 in each sequence: CBA, BAC, BCA.
Groups:
- Treatment ABC: Treatment A: Apixaban + Placebo (Saline solution): Apixaban 10 mg oral Tablet twice daily (BID) on Days 1- 3; on Day 4: Single 10 mg Dose Apixaban followed 3hours (hrs) later by Saline solution (placebo) 0 international units per kilogram of body weight (IU/kg) intravenous infusion (IV) for 30 minutes.
  Treatment B: Apixaban + Cofact [4-Factor prothrombin complex concentrate (PCC)]: Apixaban 10 mg oral Tablet BID on Days 1- 3; Day 4: Single 10 mg Dose Apixaban followed 3hrs later by Cofact (4-Factor PCC) 50 IU/kg IV infusion for 30 minutes.
  Treatment C: Apixaban + Beriplex P/N (4-Factor PCC): Apixaban 10 mg oral Tablet BID on Days 1- 3; Day 4: Single 10 mg Dose Apixaban followed 3hrs later by Beriplex P/N (4-Factor PCC) 50 IU/kg IV infusion for 30 min.
- Treatment ACB: Treatment A: Apixaban + Placebo (Saline solution): Apixaban 10 mg oral Tablet twice daily (BID)Days 1- 3; Day 4: Single 10 mg Dose Apixaban followed 3hrs later by Saline solution (placebo) 0 IU/kg IV infusion for 30 minutes.
  Treatment C: Apixaban + Beriplex P/N (4-Factor PCC): Apixaban 10 mg oral Tablet BID Days 1- 3; Day 4: Single 10 mg Dose Apixaban followed 3hrs later by Beriplex P/N (4-Factor PCC) 50 IU/kg IV infusion for 30 minutes.
  Treatment B: Apixaban + Cofact (4-Factor PCC): Apixaban 10 mg oral Tablet BID Days 1- 3; Day 4: Single 10 mg Dose Apixaban followed 3hrs later by Cofact (4-Factor PCC) 50 IU/kg IV infusion for 30 minutes.
- Treatment BAC: Treatment B: Apixaban + Cofact (4-Factor PCC): Apixaban 10 mg oral Tablet BID Days 1- 3; Day 4: Single 10 mg Dose Apixaban followed 3hrs later by Cofact (4-Factor PCC) 50 IU/kg IV infusion for 30 minutes.
  Treatment A: Apixaban + Placebo (Saline solution): Apixaban 10 mg oral Tablet twice daily (BID)Days 1- 3; Day 4: Single 10 mg Dose Apixaban followed 3hrs later by Saline solution (placebo) 0 IU/kg IV infusion for 30 minutes.
  Treatment C: Apixaban + Beriplex P/N (4-Factor PCC): Apixaban 10 mg oral Tablet BID Days 1- 3; Day 4: Single 10 mg Dose Apixaban followed 3hrs later by Beriplex P/N (4-Factor PCC) 50 IU/kg IV infusion for 30 minutes.
- Treatment BCA: Treatment B: Apixaban + Cofact (4-Factor PCC): Apixaban 10 mg oral Tablet BID Days 1- 3; Day 4: Single 10 mg Dose Apixaban followed 3hrs later by Cofact (4-Factor PCC) 50 IU/kg IV infusion for 30 minutes.
  Treatment C: Apixaban + Beriplex P/N (4-Factor PCC): Apixaban 10 mg oral Tablet BID Days 1- 3; Day 4: Single 10 mg Dose Apixaban followed 3hrs later by Beriplex P/N (4-Factor PCC) 50 IU/kg IV infusion for 30 minutes.
  Treatment A: Apixaban + Placebo (Saline solution): Apixaban 10 mg oral Tablet twice daily (BID)Days 1- 3; Day 4: Single 10 mg Dose Apixaban followed 3hrs later by Saline solution (placebo) 0 IU/kg IV infusion for 30 minutes.
- Treatment CAB: Treatment C: Apixaban + Beriplex P/N (4-Factor PCC): Apixaban 10 mg oral Tablet BID Days 1- 3; Day 4: Single 10 mg Dose Apixaban followed 3hrs later by Beriplex P/N (4-Factor PCC) 50 IU/kg IV infusion for 30 minutes.
  Treatment A: Apixaban + Placebo (Saline solution): Apixaban 10 mg oral Tablet twice daily (BID)Days 1- 3; Day 4: Single 10 mg Dose Apixaban followed 3hrs later by Saline solution (placebo) 0 IU/kg IV infusion for 30 minutes.
  Treatment B: Apixaban + Cofact (4-Factor PCC): Apixaban 10 mg oral Tablet BID Days 1- 3; Day 4: Single 10 mg Dose Apixaban followed 3hrs later by Cofact (4-Factor PCC) 50 IU/kg IV infusion for 30 minutes.
- Treatment CBA: Treatment C: Apixaban + Beriplex P/N (4-Factor PCC): Apixaban 10 mg oral Tablet BID Days 1- 3; Day 4: Single 10 mg Dose Apixaban followed 3hrs later by Beriplex P/N (4-Factor PCC) 50 IU/kg IV infusion for 30 minutes.
  Treatment B: Apixaban + Cofact (4-Factor PCC): Apixaban 10 mg oral Tablet BID Days 1- 3; Day 4: Single 10 mg Dose Apixaban followed 3hrs later by Cofact (4-Factor PCC) 50 IU/kg IV infusion for 30 minutes.
  Treatment A: Apixaban + Placebo (Saline solution): Apixaban 10 mg oral Tablet twice daily (BID)Days 1- 3; Day 4: Single 10 mg Dose Apixaban followed 3hrs later by Saline solution (placebo) 0 IU/kg IV infusion for 30 minutes.
Period: Overall Study
Arm/Group | Treatment ABC | Treatment ACB | Treatment BAC | Treatment BCA | Treatment CAB | Treatment CBA
Started | 3 | 3 | 2 | 2 | 3 | 2
Completed | 3 | 3 | 2 | 2 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study medication.
Groups:
- All Treated Participants: Treated population included all participants who received at least one dose of study medication. Participants received 10 mg apixaban BID on Days 1-3 and on Day 4 received a single dose of 10 mg apixaban followed 3 hours later by an IV infusion of 50 IU/kg prothrombin complex concentrate (PCC) (which was either Cofact or Beriplex P/N) or the participant received an IV infusion of placebo (saline solution). Participants were randomized on Day 1 to one of 6 treatment sequences (ABC, ACB, BAC, BCA, CAB and CBA). There were 3 treatment periods with a total of 3 participants in each of 3 sequences (ABC, ACB, CAB) and 2 participants in each of 3 other sequences (CBA, BAC, BCA) for a total of 15 participants who participated in this open label, randomized, crossover study.
Arm/Group | All Treated Participants
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (7.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 13
Race/Ethnicity, Customized [Number; unit: participants]
  White | 14
  Black/African American | 1
Region of Enrollment [Number; unit: participants]
  Germany | 15
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI measured as kilograms of body weight divided by meter of height, squared (kg/m^2).
  kg/m^2 | 24.5 (2.50)
Weight [Mean (Standard Deviation); unit: kilograms] | 76.5 (7.96)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacodynamic (PD) Parameter: Adjusted Mean Change in Endogenous Thrombin Potential (ETP) From Day 4 Pre-Infusion (PCC or Placebo) Baseline at Day 4, 30 Minutes Post Infusion of PCC or Placebo
Description: ETP was evaluated using a Thrombin Generation Assay (TGA), a validated automated ex vivo assay performed on platelet-poor plasma samples and based on the automated, calibrated thrombin generation method: thrombin formation was triggered with recombinant tissue factor and phospholipids. Thrombin concentration in each sample was calculated over time by measuring the cleavage of a fluorogenic substrate in the context of a paired calibration sample. Dedicated software (Thrombinoscope, Thrombinoscope B.V., Maastricht, The Netherlands) performed the calculations and derived ETP as area under the curve from the resulting "thrombogram" curve. Pre-infusion baseline= sample on Day 4, 3 hours post apixaban dose (just prior to IV infusion of PCC or placebo). Samples on Day 4 were obtained at 0 (pre-dose), 0.5, 1, 2, 3 hours post apixaban dose and at 0.5, 1, 2, 4, 6, 9, 21, 45, and 69 hours post infusion (PCC or Placebo) in each treatment period. ETP was measured as nanomolar*minute (nM*min).
Time Frame: Day 4 at 3 hours post apixaban dose and prior to infusion (Pre-infusion Baseline), Day 4 at 30 minutes post infusion (PCC or Placebo)
Population: PD Population included all participants who received any study medication and had PD data available for at least the analysis-specified baseline and 30 minutes after the start of the study drug infusion. 1 participant who received a partial PCC dose (approximately 2 IU/kg) was excluded from this summary analysis.
Measure: Mean (95% Confidence Interval); unit: nM*min
Groups:
- Treatment A: Apixaban + Placebo: Treatment A: Apixaban + Placebo (Saline solution): Apixaban 10 mg oral Tablet BID on Days 1- 3; on Day 4: Single 10 mg Dose Apixaban followed 3hours later by IV infusion of Saline solution (placebo) 0 international units per kilogram of body weight (IU/kg) for 30 minutes.
- Treatment B: Apixaban + Cofact (4-Factor PCC): Treatment B: Apixaban + Cofact (4-Factor PCC): Apixaban 10 mg oral Tablet BID on Days 1- 3; on Day 4: Single 10 mg Dose Apixaban followed 3hours later by IV infusion of Cofact (4-Factor PCC) 50 IU/kg for 30 minutes.
- Treatment C: Apixaban + Beriplex P/N (4-Factor PCC): Treatment C: Apixaban + Beriplex P/N (4-Factor PCC): Apixaban 10 mg oral Tablet BID on Days 1- 3; on Day 4: Single 10 mg Dose Apixaban followed 3hours later by IV infusion of Beriplex P/N (4-Factor PCC) 50 IU/kg for 30 minutes.
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Number analyzed (Participants) | 15 | 14 | 15
nM*min | 95.8 [21.3 to 170.2] | 521.0 [314.6 to 727.4] | 186.3 [49.7 to 322.9]
Statistical Analysis 1: Comparison: Treatment A: Apixaban + Placebo vs Treatment B: Apixaban + Cofact (4-Factor PCC); The ETP change from pre-PCC baseline was analyzed using a mixed effect model that included treatment, sequence, and period as main effects. A hierarchical analysis was conducted with comparisons beginning with the primary endpoint and continuing through secondary endpoints (ETP; TGA lag time; TGA time to peak; TGA peak; TGA velocity index; PT; INR; aPTT; AXA). If resulting p-value was < 0.05, then the next comparison of interest was made until p>0.05 at which point, comparisons ended; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; mixed effect model = 425.3, 95% CI 2-sided [219.8 to 630.7] — Treatment B versus Treatment A
Statistical Analysis 2: Comparison: Treatment A: Apixaban + Placebo vs Treatment C: Apixaban + Beriplex P/N (4-Factor PCC); ETP change from pre-PCC baseline was analyzed using mixed effect model, including treatment, sequence, and period as main effects. Hierarchical analysis was conducted with comparisons beginning with primary endpoint and continuing through secondary endpoints (ETP; TGA lag time; TGA time to peak; TGA peak; TGA velocity index; PT; INR; aPTT; AXA). If resulting p-value was < 0.05, then the next comparison of interest was made until p>0.05 at which point, comparisons ended; Test type: Superiority or Other; p = 0.131, Mixed Models Analysis — In the hierarchical analysis, no statistical inferences were drawn from the analysis results for any secondary endpoint since a non-significant treatment difference was observed for the primary endpoint; mixed effect model = 90.6, 95% CI 2-sided [-31.3 to 212.4] — Treatment C versus Treatment A

2. Secondary Outcome: PD Parameters: Adjusted Mean Change in TGA Lag Time and Adjusted Mean Change in TGA Time to Peak From Day 4 Pre-Infusion (PCC or Placebo) Baseline at Day 4, 30 Minutes Post Infusion of PCC or Placebo
Description: TGA is a validated automated ex vivo assay performed on platelet-poor plasma samples and based on the automated, calibrated thrombin generation method: thrombin formation was triggered with recombinant tissue factor and phospholipids and the concentration in each sample was calculated over time by measuring the cleavage of a fluorogenic substrate in the context of a paired calibration sample; dedicated software program was Thrombinoscope, B.V., Maastricht, The Netherlands. Samples on Day 4 were obtained at 0, 0.5, 1, 2, 3 hours post apixaban dose and at 0.5, 1, 2, 4, 6, 9, 21, 45, and 69 hours post infusion (PCC or Placebo) in each treatment period. Lag Time and Time to Peak parameters were measured in minutes.
Time Frame: Day 4 at 3 hours post apixaban dose and prior to infusion (Pre-infusion Baseline), Day 4 at 30 minutes post infusion.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Number analyzed (Participants) | 15 | 14 | 15
minutes
  TGA Lag Time (n=15, 14, 15) | -0.16 [-0.59 to 0.26] | -0.38 [-0.85 to 0.10] | -0.32 [-0.75 to 0.10]
  TGA Time to Peak (n=15, 14, 15) | -1.29 [-3.45 to 0.87] | 0.06 [-1.30 to 1.42] | 3.32 [1.97 to 4.68]
Statistical Analysis 1: Comparison: Treatment A: Apixaban + Placebo vs Treatment B: Apixaban + Cofact (4-Factor PCC); TGA Lag Time. ETP change from pre-PCC baseline was analyzed using a mixed effect model that included treatment, sequence, and period as main effects. A hierarchical analysis was conducted with comparisons beginning with the primary endpoint and continuing through secondary endpoints (ETP; TGA lag time; TGA time to peak; TGA peak; TGA velocity index; PT; INR; aPTT; AXA). If resulting p-value was < 0.05, then the next comparison of interest was made until p>0.05 at which point, comparisons ended; Test type: Superiority or Other; p = 0.389, Mixed Models Analysis — In the hierarchical analysis, no statistical inferences were drawn from the analysis results for other secondary endpoints since a non-significant treatment difference was observed for this first secondary endpoint (TGA lag time); mixed effect model = -0.21, 95% CI 2-sided [-0.73 to 0.30] — Treatment B versus Treatment A
Statistical Analysis 2: Comparison: Treatment A: Apixaban + Placebo vs Treatment C: Apixaban + Beriplex P/N (4-Factor PCC); Lag Time. ETP change from pre-PCC baseline was analyzed using mixed effect model, including treatment, sequence, and period as main effects. Hierarchical analysis was conducted with comparisons beginning with primary endpoint and continuing through secondary endpoints (ETP; TGA lag time; TGA time to peak; TGA peak; TGA velocity index; PT; INR; aPTT; AXA). If resulting p-value was < 0.05, then the next comparison of interest was made until p>0.05 at which point, comparisons ended; Test type: Superiority or Other; p = 0.142, Mixed Models Analysis — In the hierarchical analysis, no statistical inferences were drawn from the analysis results for this secondary endpoint since a non-significant treatment difference was observed for the primary endpoint; mixed effect model = -0.16, 95% CI 2-sided [-0.38 to 0.06] — Treatment C versus Treatment A
Statistical Analysis 3: Comparison: Treatment A: Apixaban + Placebo vs Treatment B: Apixaban + Cofact (4-Factor PCC); Time to Peak. ETP change from pre-PCC baseline was analyzed using a mixed effect model that included treatment, sequence, and period as main effects. A hierarchical analysis was conducted with comparisons beginning with the primary endpoint and continuing through secondary endpoints (ETP; TGA lag time; TGA time to peak; TGA peak; TGA velocity index; PT; INR; aPTT; AXA). If resulting p-value was < 0.05, then the next comparison of interest was made until p>0.05 at which point, comparisons ended; Test type: Superiority or Other; p = 0.200, Mixed Models Analysis — In the hierarchical analysis, no statistical inferences were drawn from the analysis results for this secondary endpoint since a non-significant treatment difference was observed for the first secondary endpoint (TGA lag time); mixed effect model = 1.35, 95% CI 2-sided [-0.81 to 3.52] — Treatment B versus Treatment A
Statistical Analysis 4: Comparison: Treatment A: Apixaban + Placebo vs Treatment C: Apixaban + Beriplex P/N (4-Factor PCC); Time to Peak. ETP change from pre-PCC baseline was analyzed using mixed effect model, including treatment, sequence, and period as main effects. Hierarchical analysis was conducted with comparisons beginning with primary endpoint and continuing through secondary endpoints (ETP; TGA lag time; TGA time to peak; TGA peak; TGA velocity index; PT; INR; aPTT; AXA). If resulting p-value was < 0.05, then the next comparison of interest was made until p>0.05 at which point, comparisons ended; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 2]; mixed effect model = 4.62, 95% CI 2-sided [2.80 to 6.44] — Treatment C versus Treatment A

3. Secondary Outcome: PD Parameter: Adjusted Mean Change in TGA Peak Height From Day 4 Pre-Infusion (PCC or Placebo) Baseline at Day 4, 30 Minutes Post Infusion of PCC or Placebo
Description: TGA is a validated automated ex vivo assay performed on platelet-poor plasma samples and based on the automated, calibrated thrombin generation method: thrombin formation was triggered with recombinant tissue factor and phospholipids and the concentration in each sample was calculated over time by measuring the cleavage of a fluorogenic substrate in the context of a paired calibration sample; dedicated software program was Thrombinoscope, B.V., Maastricht, The Netherlands. Samples on Day 4 were obtained at 0, 0.5, 1, 2, 3 hours post apixaban dose and at 0.5, 1, 2, 4, 6, 9, 21, 45, and 69 hours post infusion (PCC or Placebo) in each treatment period. Peak height parameter was measured in nanomolar (nM).
Time Frame: Day 4 at 3 hours post apixaban dose and prior to infusion (Pre-infusion Baseline), Day 4 at 30 minutes post infusion.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: nM
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Number analyzed (Participants) | 15 | 14 | 15
nM | 11.1 [5.1 to 17.0] | 32.1 [15.2 to 49.1] | 4.7 [-3.3 to 12.7]
Statistical Analysis 1: Comparison: Treatment A: Apixaban + Placebo vs Treatment B: Apixaban + Cofact (4-Factor PCC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.014, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 3]; mixed effect model = 21.1, 95% CI 2-sided [4.9 to 37.2] — Treatment B versus Treatment A
Statistical Analysis 2: Comparison: Treatment A: Apixaban + Placebo vs Treatment C: Apixaban + Beriplex P/N (4-Factor PCC); [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.076, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 2]; mixed effect model = -6.4, 95% CI 2-sided [-13.5 to 0.8] — Treatment C versus Treatment A

4. Secondary Outcome: PD Parameter: Adjusted Mean Change in TGA Velocity Index From Day 4 Pre-Infusion (PCC or Placebo) Baseline at Day 4, 30 Minutes Post Infusion of PCC or Placebo
Description: TGA is a validated automated ex vivo assay performed on platelet-poor plasma samples and based on the automated, calibrated thrombin generation method: thrombin formation was triggered with recombinant tissue factor and phospholipids and the concentration in each sample was calculated over time by measuring the cleavage of a fluorogenic substrate in the context of a paired calibration sample; dedicated software program was Thrombinoscope, B.V., Maastricht, The Netherlands. Samples on Day 4 were obtained at 0, 0.5, 1, 2, 3 hours post apixaban dose and at 0.5, 1, 2, 4, 6, 9, 21, 45, and 69 hours post infusion (PCC or Placebo) in each treatment period. TGA Velocity Index parameter was measured in nM per minute (nM/min).
Time Frame: Day 4 at 3 hours post apixaban dose and prior to infusion (Pre-infusion Baseline), Day 4 at 30 minutes post infusion.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: nM/min
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Number analyzed (Participants) | 15 | 14 | 15
nM/min | 3.4 [-0.5 to 7.3] | 3.4 [-1.5 to 8.2] | -3.2 [-5.4 to -0.9]
Statistical Analysis 1: Comparison: Treatment A: Apixaban + Placebo vs Treatment B: Apixaban + Cofact (4-Factor PCC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.996, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 3]; mixed effect model = 0.0, 95% CI 2-sided [-5.6 to 5.6] — Treatment B versus Treatment A
Statistical Analysis 2: Comparison: Treatment A: Apixaban + Placebo vs Treatment C: Apixaban + Beriplex P/N (4-Factor PCC); [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 2]; mixed effect model = -6.5, 95% CI 2-sided [-9.5 to -3.6] — Treatment C versus Treatment A

5. Secondary Outcome: PD Parameter: Adjusted Mean Change in Coagulation Parameters Prothrombin Time (PT) and Activated Partial Thromboplastin Time (aPTT) From Day 4 Pre-Infusion (PCC or Placebo) Baseline at Day 4, 30 Minutes Post Infusion of PCC or Placebo
Description: Coagulation parameters were evaluated by Quintiles Laboratories Europe using an ACL TOP analyzer and Instrumentation Laboratory reagents [HemosIL(Registered) Recombiplastin 2G for PT and Synthasil for aPTT]. A second PT was also measured at Esoterix using a Diagnostica Stago STA Compact coagulation analyzer and Diagnostica Stago reagents STA-Neoplastin CI Plus (Registered). Samples on Day 4 were obtained at 0 and 3 hours post apixaban dose and at 0.5, 1, 2, 4, 6, 9, 21, 45, and 69 hours post infusion (PCC or Placebo) in each treatment period. PT (Neoplastin CT+), PT (Recombiplastin 2G) and activated partial thromboplastin time (aPTT) parameters were measured in seconds.
Time Frame: Day 4 at 3 hours post apixaban dose and prior to infusion (Pre-infusion Baseline), Day 4 at 30 minutes post infusion.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Number analyzed (Participants) | 15 | 14 | 15
seconds
  PT (Neoplastin CI+) (n=15, 14, 15) | -0.21 [-0.44 to 0.02] | -1.85 [-2.30 to -1.40] | -1.68 [-1.99 to -1.38]
  PT (Recombiplastin 2G) (n=15, 14, 15) | 0.35 [-0.13 to 0.83] | -2.24 [-2.74 to -1.75] | -1.54 [-2.16 to -0.92]
  aPTT (n=15, 14, 15) | 1.13 [0.38 to 1.87] | 9.60 [7.69 to 11.51] | 3.43 [2.66 to 4.20]
Statistical Analysis 1: Comparison: Treatment A: Apixaban + Placebo vs Treatment B: Apixaban + Cofact (4-Factor PCC); PT (Neoplastin CI+). ETP change from pre-PCC baseline was analyzed using mixed effect model that included treatment, sequence, and period as main effects. Hierarchical analysis was conducted with comparisons beginning with primary endpoint and continuing through secondary endpoints (ETP; TGA lag time; TGA time to peak; TGA peak; TGA velocity index; PT; INR; aPTT; AXA). If resulting p-value was < 0.05, then the next comparison of interest was made until p>0.05 at which point, comparisons ended; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 3]; mixed effect model = -1.64, 95% CI 2-sided [-2.16 to -1.12] — Treatment B versus Treatment A
Statistical Analysis 2: Comparison: Treatment A: Apixaban + Placebo vs Treatment C: Apixaban + Beriplex P/N (4-Factor PCC); PT (Neoplastin CI+). ETP change from pre-PCC baseline was analyzed using mixed effect model, including treatment, sequence, and period as main effects. Hierarchical analysis was conducted with comparisons beginning with primary endpoint and continuing through secondary endpoints (ETP; TGA lag time; TGA time to peak; TGA peak; TGA velocity index; PT; INR; aPTT; AXA). If resulting p-value was < 0.05, then the next comparison of interest was made until p>0.05 at which point, comparisons ended; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 2]; mixed effect model = -1.47, 95% CI 2-sided [-1.95 to -0.99] — Treatment C versus Treatment A
Statistical Analysis 3: Comparison: Treatment A: Apixaban + Placebo vs Treatment B: Apixaban + Cofact (4-Factor PCC); PT (Recombiplastin 2G). ETP change from pre-PCC baseline was analyzed using mixed effect model, including treatment, sequence, and period as main effects. Hierarchical analysis was conducted with comparisons beginning with primary endpoint and continuing through secondary endpoints (ETP; TGA lag time; TGA time to peak; TGA peak; TGA velocity index; PT; INR; aPTT; AXA). If resulting p-value was < 0.05, then the next comparison of interest was made until p>0.05 at which point, comparisons ended; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 3]; mixed effect model = -2.59, 95% CI 2-sided [-3.30 to -1.89] — Treatment B versus Treatment A
Statistical Analysis 4: Comparison: Treatment A: Apixaban + Placebo vs Treatment C: Apixaban + Beriplex P/N (4-Factor PCC); [analysis description as in outcome 5, analysis 3]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 2]; mixed effect model = -1.89, 95% CI 2-sided [-2.59 to -1.20] — Treatment C versus Treatment A
Statistical Analysis 5: Comparison: Treatment A: Apixaban + Placebo vs Treatment B: Apixaban + Cofact (4-Factor PCC); aPTT. The ETP change from pre-PCC baseline was analyzed using a mixed effect model and included treatment, sequence, and period as main effects. Hierarchical analysis was conducted with comparisons beginning with primary endpoint and continuing through secondary endpoints (ETP; TGA lag time; TGA time to peak; TGA peak; TGA velocity index; PT; INR; aPTT; AXA). If resulting p-value was < 0.05, then the next comparison of interest was made until p>0.05 at which point, comparisons ended; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 3]; mixed effect model = 8.47, 95% CI 2-sided [6.29 to 10.66] — Treatment B versus Treatment A
Statistical Analysis 6: Comparison: Treatment A: Apixaban + Placebo vs Treatment C: Apixaban + Beriplex P/N (4-Factor PCC); aPTT. ETP change from pre-PCC baseline was analyzed using mixed effect model, including treatment, sequence, and period as main effects. Hierarchical analysis was conducted with comparisons beginning with primary endpoint and continuing through secondary endpoints (ETP; TGA lag time; TGA time to peak; TGA peak; TGA velocity index; PT; INR; aPTT; AXA). If resulting p-value was < 0.05, then the next comparison of interest was made until p>0.05 at which point, comparisons ended; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 2]; mixed effect model = 2.30, 95% CI 2-sided [1.28 to 3.32] — Treatment C versus Treatment A

6. Secondary Outcome: PD Parameter: Adjusted Mean Change in Coagulation Parameter International Normalized Ratio (INR) From Day 4 Pre-Infusion (PCC or Placebo) Baseline at Day 4, 30 Minutes Post Infusion of PCC or Placebo
Description: Coagulation parameters were evaluated by Quintiles Laboratories Europe using an ACL TOP analyzer and Instrumentation Laboratory reagents [HemosIL(Registered) Recombiplastin 2G for PT and Synthasil for aPTT]. A second PT was also measured at Esoterix using a Diagnostica Stago STA Compact coagulation analyzer and Diagnostica Stago reagents STA-Neoplastin CI Plus (Registered). Samples on Day 4 were obtained at 0 and 3 hours post apixaban dose and at 0.5, 1, 2, 4, 6, 9, 21, 45, and 69 hours post infusion (PCC or Placebo) in each treatment period. INR was measured as a fraction.
Time Frame: Day 4 at 3 hours post apixaban dose and prior to infusion (Pre-infusion Baseline), Day 4 at 30 minutes post infusion.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: fraction
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Number analyzed (Participants) | 15 | 14 | 15
fraction
  INR (Neoplastin CI+) (n=15, 14, 15) | -0.015 [-0.048 to 0.019] | -0.213 [-0.274 to -0.152] | -0.185 [-0.218 to -0.152]
  INR (Recombiplastin 2G) (n=15, 14, 15) | 0.032 [-0.014 to 0.077] | -0.207 [-0.254 to -0.161] | -0.144 [-0.202 to -0.086]
Statistical Analysis 1: Comparison: Treatment A: Apixaban + Placebo vs Treatment B: Apixaban + Cofact (4-Factor PCC); INR (Neoplastin CI+). ETP change from pre-PCC baseline was analyzed using mixed effect model, including treatment, sequence, and period as main effects. Hierarchical analysis was conducted with comparisons beginning with primary endpoint and continuing through secondary endpoints (ETP; TGA lag time; TGA time to peak; TGA peak; TGA velocity index; PT; INR; aPTT; AXA). If resulting p-value was < 0.05, then the next comparison of interest was made until p>0.05 at which point, comparisons ended; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 3]; mixed effect model = -0.198, 95% CI 2-sided [-0.266 to -0.130] — Treatment B versus Treatment A
Statistical Analysis 2: Comparison: Treatment A: Apixaban + Placebo vs Treatment C: Apixaban + Beriplex P/N (4-Factor PCC); [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 2]; mixed effect model = -0.170, 95% CI 2-sided [-0.229 to -0.111] — Treatment C versus Treatment A
Statistical Analysis 3: Comparison: Treatment A: Apixaban + Placebo vs Treatment B: Apixaban + Cofact (4-Factor PCC); INR (Recombiplastin 2G). ETP change from pre-PCC baseline was analyzed using mixed effect model, including treatment, sequence, and period as main effects. Hierarchical analysis was conducted with comparisons beginning with primary endpoint and continuing through secondary endpoints (ETP; TGA lag time; TGA time to peak; TGA peak; TGA velocity index; PT; INR; aPTT; AXA). If resulting p-value was < 0.05, then the next comparison of interest was made until p>0.05 at which point, comparisons ended; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 3]; mixed effect model = -0.239, 95% CI 2-sided [-0.305 to -0.173] — Treatment B versus Treatment A
Statistical Analysis 4: Comparison: Treatment A: Apixaban + Placebo vs Treatment C: Apixaban + Beriplex P/N (4-Factor PCC); [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 2]; mixed effect model = -0.176, 95% CI 2-sided [-0.242 to -0.110] — Treatment C versus Treatment A

7. Secondary Outcome: PD Parameter: Adjusted Mean Change in Plasma Anti-Xa Activity From Day 4 Pre-Infusion (PCC or Placebo) Baseline at Day 4, 30 Minutes Post Infusion of PCC or Placebo
Description: Anti-FXa activity was measured using a validated method at Esoterix Coagulation Laboratory (Englewood, CO) using the Diagnostica Stago Rotachrom (Registered) Heparin assay on a STA-Compact (Registered) analyzer. Samples on Day 4 were obtained at 0, 0.5, 1, 2, 3 hours post apixaban dose and at 0.5, 1, 2, 4, 6, 9, 21, 45, and 69 hours post infusion (PCC or Placebo) in each treatment period. The results of this chromogenic assay were reported in low molecular weight heparin (LMWH) activity units per milliliter (U/mL), which are equivalent to international units per milliliter (IU/mL) with assay reportable range: 0.1 to 18.4 IU/mL.
Time Frame: Day 4 at 3 hours post apixaban dose and prior to infusion (Pre-infusion Baseline), Day 4 at 30 minutes post infusion.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Number analyzed (Participants) | 15 | 14 | 15
U/mL | -0.368 [-0.588 to -0.148] | -0.607 [-0.827 to -0.387] | -0.538 [-0.683 to -0.393]
Statistical Analysis 1: Comparison: Treatment A: Apixaban + Placebo vs Treatment B: Apixaban + Cofact (4-Factor PCC); Anti-Xa Activity. ETP change from pre-PCC baseline was analyzed using mixed effect model, including treatment, sequence, and period as main effects. Hierarchical analysis was conducted with comparisons beginning with primary endpoint and continuing through secondary endpoints (ETP; TGA lag time; TGA time to peak; TGA peak; TGA velocity index; PT; INR; aPTT; AXA). If resulting p-value was < 0.05, then the next comparison of interest was made until p>0.05 at which point, comparisons ended; Test type: Superiority or Other; p = 0.204, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 3]; mixed effect models = -0.239, 95% CI 2-sided [-0.625 to 0.146] — Treatment B versus Treatment A
Statistical Analysis 2: Comparison: Treatment A: Apixaban + Placebo vs Treatment C: Apixaban + Beriplex P/N (4-Factor PCC); [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.114, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 2]; mixed effect models = -0.170, 95% CI 2-sided [-0.389 to 0.048] — Treatment C versus Treatment A

8. Secondary Outcome: PD Parameter: Adjusted Mean Change in TGA Lag Time and TGA Time to Peak From Day 1 Pre-Dose Apixaban Baseline at Day 4, 30 Minutes Post Infusion of PCC or Placebo
Description: TGA is a validated, automated ex vivo assay performed on platelet-poor plasma samples and based on the automated, calibrated thrombin generation method: thrombin formation was triggered with recombinant tissue factor and phospholipids and the concentration in each sample was calculated over time by measuring the cleavage of a fluorogenic substrate in the context of a paired calibration sample; dedicated software program was Thrombinoscope, B.V., Maastricht, The Netherlands. Baseline was Day 1, 0 hour pre-dose apixaban. Samples on Day 4 were obtained at 0, 0.5, 1, 2, 3 hours post apixaban dose and 0.5, 1, 2, 4, 6, 9, 21, 45, and 69 hours post infusion (PCC or Placebo) in each treatment period. TGA Lag Time and Time to Peak parameters were measured in minutes.
Time Frame: Day 1, pre-dose apixaban (Baseline), Day 4, 30 minutes post infusion.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Number analyzed (Participants) | 15 | 14 | 15
minutes
  TGA Lag Time (n=15,14,15) | 3.56 [3.16 to 3.96] | 3.36 [2.86 to 3.86] | 3.40 [3.05 to 3.76]
  TGA Time to Peak (n=15,14,15) | 6.42 [3.96 to 8.89] | 7.90 [6.41 to 9.40] | 10.81 [9.22 to 12.39]

9. Secondary Outcome: PD Parameter: Adjusted Mean Change in TGA Peak Height From Day 1 Pre-Dose Apixaban Baseline at Day 4, 30 Minutes Post Infusion of PCC or Placebo
Description: as for outcome 8
Time Frame: Day 1, pre-dose apixaban (Baseline), Day 4, 30 minutes post infusion.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: nM
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Number analyzed (Participants) | 15 | 14 | 15
nM | -196.1 [-205.6 to -186.6] | -174.9 [-192.3 to -157.5] | -202.7 [-211.7 to -193.7]

10. Secondary Outcome: PD Parameter: Adjusted Mean Change in TGA Velocity Index From Day 1 Pre-Dose Apixaban Baseline at Day 4, 30 Minutes Post Infusion of PCC or Placebo
Description: TGA is a validated, automated ex vivo assay performed on platelet-poor plasma samples and based on the automated, calibrated thrombin generation method: thrombin formation was triggered with recombinant tissue factor and phospholipids and the concentration in each sample was calculated over time by measuring the cleavage of a fluorogenic substrate in the context of a paired calibration sample; dedicated software program was Thrombinoscope, B.V., Maastricht, The Netherlands. Baseline was Day 1, 0 hour (pre-dose apixaban). Samples on Day 4 were obtained at 0, 0.5, 1, 2, 3 hours post apixaban dose and at 0.5, 1, 2, 4, 6, 9, 21, 45, and 69 hours post infusion (PCC or Placebo) in each treatment period. TGA velocity index was measured in nM/min.
Time Frame: Day 1, pre-dose apixaban (Baseline), Day 4, 30 minutes post infusion.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: nM/min
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Number analyzed (Participants) | 15 | 14 | 15
nM/min | -63.7 [-67.1 to -60.3] | -63.6 [-68.3 to -58.9] | -71.5 [-74.1 to -69.0]

11. Primary Outcome: PD Parameter: Adjusted Mean Change in Endogenous Thrombin Potential (ETP) From Day 1 Pre-Dose Apixaban Baseline at Day 4, 30 Minutes Post Infusion of PCC or Placebo
Description: ETP was evaluated using a Thrombin Generation Assay (TGA), a validated automated ex vivo assay performed on platelet-poor plasma samples and based on the automated, calibrated thrombin generation method: thrombin formation was triggered with recombinant tissue factor and phospholipids. Thrombin concentration in each sample was calculated over time by measuring the cleavage of a fluorogenic substrate in the context of a paired calibration sample. A dedicated software program (Thrombinoscope, Thrombinoscope B.V., Maastricht, The Netherlands) performed the calculations and derived ETP as area under the curve from the resulting "thrombogram" curve. Pre-dose Apixaban baseline was Day 1 pre-dose (0 hour). Samples on Day 4 were obtained at 0, 0.5, 1, 2, 3 hours post apixaban dose and at 0.5, 1, 2, 4, 6, 9, 21, 45, and 69 hours post infusion (PCC or Placebo) in each treatment period.
Time Frame: Day 1 pre-dose apixaban (pre-apixaban Baseline), Day 4 at 30 minutes post infusion (PCC or Placebo)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: nM*minute
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Number analyzed (Participants) | 15 | 14 | 15
nM*minute | -708.0 [-791.1 to -625.0] | -276.3 [-465.8 to -86.9] | -607.7 [-701.2 to -514.2]

12. Secondary Outcome: PD Parameter: Adjusted Mean Change in Coagulation Parameters PT and aPTT From Day 1 Pre-Dose Apixaban Baseline at Day 4, 30 Minutes Post Infusion of PCC or Placebo
Description: Coagulation parameters were evaluated by Quintiles Laboratories Europe using an ACL TOP analyzer and Instrumentation Laboratory reagents [HemosIL(Registered) Recombiplastin 2G for PT and Synthasil for aPTT]. A second PT was also measured at Esoterix using a Diagnostica Stago STA Compact coagulation analyzer and Diagnostica Stago reagents STA-Neoplastin CI Plus (Registered). Baseline was Day 1, pre-apixaban dose. Samples on Day 4 were obtained at 0 and 3 hours post apixaban dose and at 0.5, 1, 2, 4, 6, 9, 21, 45, and 69 hours post infusion (PCC or Placebo) in each treatment period.
Time Frame: Day 1, pre-dose apixaban (Baseline), Day 4, 30 minutes post infusion.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Number analyzed (Participants) | 15 | 14 | 15
seconds
  PT (Neoplastin CI+) (n=15,14,15) | 2.74 [2.54 to 2.94] | 1.17 [0.65 to 1.70] | 1.31 [0.94 to 1.67]
  PT (Recombiplastin 2G) (n=15,14,15) | 4.94 [4.57 to 5.33] | 2.30 [1.74 to 2.86] | 3.01 [2.43 to 3.59]
  aPTT (n=15, 14, 15) | 7.49 [6.75 to 8.23] | 15.87 [13.91 to 17.82] | 9.68 [8.84 to 10.52]

13. Secondary Outcome: PD Parameter: Adjusted Mean Change in Coagulation Parameter INR From Day 1 Pre-Dose Apixaban Baseline at Day 4, 30 Minutes Post Infusion of PCC or Placebo
Description: Coagulation parameters were evaluated by Quintiles Laboratories Europe using an ACL TOP analyzer and Instrumentation Laboratory reagents [HemosIL(Registered) Recombiplastin 2G for PT and Synthasil for aPTT]. A second PT was also measured at Esoterix using a Diagnostica Stago STA Compact coagulation analyzer and Diagnostica Stago reagents STA-Neoplastin CI Plus (Registered). Baseline was Day 1, 0 hour pre-dose apixaban. Samples on Day 4 were obtained at 0 and 3 hours post apixaban dose and at 0.5, 1, 2, 4, 6, 9, 21, 45, and 69 hours post infusion (PCC or Placebo) in each treatment period. INR was measured as a fraction
Time Frame: Day 1, pre-dose apixaban (Baseline), Day 4, 30 minutes post infusion.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: fraction
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Number analyzed (Participants) | 15 | 14 | 15
fraction
  INR (Neoplastin CI+) (n=15,14,15) | 0.290 [0.260 to 0.321] | 0.103 [0.026 to 0.180] | 0.130 [0.084 to 0.176]
  INR (Recombiplastin 2G) (n=15,14,15) | 0.460 [0.424 to 0.497] | 0.216 [0.164 to 0.269] | 0.281 [0.227 to 0.335]

14. Secondary Outcome: Geometric Mean Maximum Observed Plasma Concentration (Cmax) of Apixaban on Day 4
Description: Plasma samples for pharmacokinetic (PK) analysis were obtained on Day 4 at 0 hour (pre-dose), 0.5, 1, 2, and 3 hours post apixaban dose, and at 0.5, 1, 2, 4, 6, 9 hours post infusion (PCC or Placebo), and at 21, 45, and 69 hours post infusion (Days 5, 6, and 7) in each treatment period. PK parameters were derived from plasma concentration versus time. Concentration of apixaban was determined using a validated liquid chromatography tandem mass spectrometry (LC/MS/MS) assay within the period of known analyte stability. Cmax was measured in nanograms per milliliter (ng/mL).
Time Frame: Day 4
Population: Those participants who received any study medication and had adequate PK profiles were included; 1 participant who received a partial PCC dose (approximately 2 IU/kg) was excluded from this summary analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Number analyzed (Participants) | 15 | 14 | 15
ng/mL | 291 (23) | 310 (29) | 290 (28)

15. Secondary Outcome: Geometric Mean Time of Maximum Observed Plasma Concentration (Tmax) of Apixaban on Day 4
Description: Plasma samples for PK analysis were obtained on Day 4 at 0 hour (pre-dose), 0.5, 1, 2, and 3 hours post apixaban dose, and at 0.5, 1, 2, 4, 6, 9 hours post infusion (PCC or Placebo), and at 21, 45, and 69 hours post infusion (Days 5, 6, and 7) in each treatment period. PK parameters were derived from plasma concentration versus time. Concentration of apixaban was determined using a validated LC/MS/MS assay within the period of known analyte stability. Tmax was measured in hours.
Time Frame: Day 4
Population: as for outcome 14
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Number analyzed (Participants) | 15 | 14 | 15
hours | 2.00 [1.02 to 2.98] | 2.00 [0.980 to 2.98] | 2.00 [1.00 to 2.98]

16. Secondary Outcome: Geometric Mean Area Under the Plasma Concentration-Time Curve in One Dosing Interval [AUC(0-12)] of Apixaban on Day 4
Description: Plasma samples for PK analysis were obtained on Day 4 at 0 hour (pre-dose), 0.5, 1, 2, and 3 hours post apixaban dose, and at 0.5, 1, 2, 4, 6, 9 hours post infusion (PCC or Placebo), and at 21, 45, and 69 hours post infusion (Days 5, 6, and 7) in each treatment period. PK parameters were derived from plasma concentration versus time. Concentration of apixaban was determined using a validated LC/MS/MS assay within the period of known analyte stability. AUC(0-12) was measured in ng*hours/mL (ng*h/mL)
Time Frame: Day 4
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Number analyzed (Participants) | 15 | 14 | 15
ng*h/mL | 1965 (22) | 2046 (26) | 2010 (26)

17. Secondary Outcome: Adjusted Geometric Mean AUC (0-12) of Apixaban on Day 4
Description: Plasma samples for PK analysis were obtained on Day 4 at 0 hour (pre-dose), 0.5, 1, 2, and 3 hours post apixaban dose, and at 0.5, 1, 2, 4, 6, 9 hours post infusion (PCC or Placebo), and at 21, 45, and 69 hours post infusion (Days 5, 6, and 7) in each treatment period. PK parameters were derived from plasma concentration versus time. Concentration of apixaban was determined using a validated LC/MS/MS assay within the period of known analyte stability.
Time Frame: Day 4
Population: as for outcome 14
Measure: Geometric Mean (90% Confidence Interval); unit: ng*h/mL
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Number analyzed (Participants) | 15 | 14 | 15
ng*h/mL | 1972 [1752 to 2219] | 2049 [1818 to 2309] | 2014 [1809 to 2241]
Statistical Analysis 1: Comparison: Treatment A: Apixaban + Placebo vs Treatment B: Apixaban + Cofact (4-Factor PCC); Analysis used a linear mixed effect model including treatment, period, and sequence as fixed effects and within-participant measurements as repeated measures. Point estimates and 90% confidence intervals (CIs) for differences on the log scale were exponentiated to obtain estimates for ratios of geometric means on the original scale between each PCC treatment and placebo (ie, Treatment B versus Treatment A, and Treatment C versus Treatment A). No adjustment was made for multiplicity; Test type: Superiority or Other; mixed effect model = 1.039, 90% CI 2-sided [0.972 to 1.111] — Treatment B versus Treatment A
Statistical Analysis 2: Comparison: Treatment A: Apixaban + Placebo vs Treatment C: Apixaban + Beriplex P/N (4-Factor PCC); Analysis used a linear mixed effect model including treatment, period, and sequence as fixed effects and within-participant measurements as repeated measures. Point estimates and 90% confidence intervals (CIs) for differences on the log scale were exponentiated to obtain estimates for ratios of geometric means on the original scale between each PCC treatment and placebo (ie, Treatment C versus Treatment A). No adjustment was made for multiplicity; Test type: Superiority or Other; mixed effect model = 1.021, 90% CI 2-sided [0.938 to 1.112] — Treatment C versus Treatment A

18. Secondary Outcome: Geometric Mean Area Under the Plasma Concentration-Time Curve From Time Zero to 24 Hours After Dose Administration [AUC(0-24)] of Apixaban on Day 4
Description: Plasma samples for PK analysis were obtained on Day 4 at 0 hour (pre-dose), 0.5, 1, 2, and 3 hours post apixaban dose, and at 0.5, 1, 2, 4, 6, 9 hours post infusion (PCC or Placebo), and at 21, 45, and 69 hours post infusion (Days 5, 6, and 7) in each treatment period. PK parameters were derived from plasma concentration versus time. Concentration of apixaban was determined using a validated LC/MS/MS assay within the period of known analyte stability. AUC(0-24) was measured in ng*h/mL.
Time Frame: Day 4
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Number analyzed (Participants) | 15 | 14 | 15
ng*h/mL | 2537 (23) | 2583 (27) | 2585 (28)

19. Secondary Outcome: Adjusted Geometric Mean AUC (0-24) for Apixaban on Day 4
Description: as for outcome 17
Time Frame: Day 4
Population: as for outcome 14
Measure: Geometric Mean (90% Confidence Interval); unit: ng*h/mL
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Number analyzed (Participants) | 15 | 14 | 15
ng*h/mL | 2546 [2258 to 2871] | 2594 [2295 to 2932] | 2592 [2315 to 2902]
Statistical Analysis 1: Comparison: Treatment A: Apixaban + Placebo vs Treatment B: Apixaban + Cofact (4-Factor PCC); Analysis used a linear mixed effect model including treatment, period, and sequence as fixed effects and within-participant measurements as repeated measures. Point estimates and 90% confidence intervals (CIs) for differences on the log scale were exponentiated to obtain estimates for ratios of geometric means on the original scale between each PCC treatment and placebo (ie, Treatment B versus Treatment A). No adjustment was made for multiplicity; Test type: Superiority or Other; mixed effect model = 1.019, 90% CI 2-sided [0.955 to 1.087] — Treatment B versus Treatment A
Statistical Analysis 2: Comparison: Treatment A: Apixaban + Placebo vs Treatment C: Apixaban + Beriplex P/N (4-Factor PCC); [analysis description as in outcome 17, analysis 2]; Test type: Superiority or Other; mixed effect model = 1.018, 90% CI 2-sided [0.940 to 1.102] — Treatment C versus Treatment A

20. Secondary Outcome: Geometric Mean Trough Observed Plasma Concentration at the End of One Dosing Interval (12h) [Cmin] of Apixaban on Day 4
Description: Plasma samples for PK analysis were obtained on Day 4 at 0 hour (pre-dose), 0.5, 1, 2, and 3 hours post apixaban dose, and at 0.5, 1, 2, 4, 6, 9 hours post infusion (PCC or Placebo), and at 21, 45, and 69 hours post infusion (Days 5, 6, and 7) in each treatment period. PK parameters were derived from plasma concentration versus time. Concentration of apixaban was determined using a validated LC/MS/MS assay within the period of known analyte stability. Cmin was measured in nanograms per milliliter (ng/mL).
Time Frame: Day 4
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Number analyzed (Participants) | 15 | 14 | 15
ng/mL | 86.0 (26) | 93.7 (37) | 95.5 (39)

21. Secondary Outcome: Mean Terminal Elimination Half-Life (T-HALF) of Apixaban on Day 4
Description: Plasma samples for PK analysis were obtained on Day 4 at 0 hour (pre-dose), 0.5, 1, 2, and 3 hours post apixaban dose, and at 0.5, 1, 2, 4, 6, 9 hours post infusion (PCC or Placebo), and at 21, 45, and 69 hours post infusion (Days 5, 6, and 7) in each treatment period. PK parameters were derived from plasma concentration versus time. Concentration of apixaban was determined using a validated LC/MS/MS assay within the period of known analyte stability. T-HALF was measured in hours
Time Frame: Day 4
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Number analyzed (Participants) | 15 | 14 | 15
hours | 10.9 (2.49) | 10.8 (2.95) | 11.0 (1.87)

22. Secondary Outcome: Number of Participants With Death, Serious Adverse Events (SAEs), Adverse Events (AEs), and Discontinuation Due to AEs - Treatment Population
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or missing relationship to study drug. Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4= Potentially Life-threatening or disabling. Medical Dictionary for Regulatory Activities (MedDRA) version 17.0 was used.
Time Frame: Day 1 to 30 days Post Last Dose
Population: Treated population: All participants who received at least one dose of study medication were analyzed.
Measure: Number; unit: participants
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Number analyzed (Participants) | 15 | 15 | 15
participants
  Adverse Events | 1 | 5 | 2
  SAEs | 0 | 0 | 0
  Discontinuation due to AEs | 0 | 0 | 0
  Death | 0 | 0 | 0

23. Secondary Outcome: Number of Participants With Marked Abnormalities (MA) in Laboratory Tests - Treated Population
Description: Blood, urine samples obtained at screening, Days -1, 4, and 7 of each treatment period, and study discharge (Day 11 of Treatment Period 3). MA: Leukocyte White Blood Cells (WBC) *10^3 cells per microliter (c/µL); High (H): > 1.2*upper limits normal (ULN) if lower limits normal (LLN) <= pre-therapy (PreRx) <= ULN; > 1.2*ULN if PreRx = Missing; > 1.5*PreRx if PreRx > ULN; > ULN if PreRx < LLN. Alanine Aminotransferase (ALT) units per liter (U/L); H: > 1.25*PreRx if PreRx > ULN; > 1.25*ULN if PreRx <= ULN; > 1.25*ULN if PreRx = Missing. Total and Direct Bilirubin in milligrams/deciliter (mg/dL) H: > 1.1*ULN if PreRx <= ULN;> 1.1*ULN if PreRx = Missing; > 1.25*PreRx if PreRx > ULN. Blood in Urine H: >= 2*PreRx if PreRx >= 1; >= 2 if PreRx < 1; >= 2 if PreRx = Missing. Urine Red Blood Cells (RBC) and Urine WBC/ high powered field (hpf) H: >= 2 if PreRx = Missing; >= 2 if PreRx < 2; >= 4 if PreRx >= 2. Crossover study: same participant with MA could be reported in multiple arms.
Time Frame: Day 1 (first dose) to Day of Study Discharge (Day 11 of Treatment Period 3)
Population: All participants who received any study medication and had available laboratory test data were analyzed. n=number of participants evaluated.
Measure: Number; unit: participants
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Number analyzed (Participants) | 15 | 15 | 15
participants
  Leukocytes High (n=15,15,15) | 0 | 1 | 0
  ALT High (n=15,15,15) | 1 | 1 | 0
  Bilirubin Direct High (n=4,4,4) | 2 | 2 | 2
  Bilirubin Total High (n=15,15,15) | 2 | 1 | 2
  Blood in Urine (n=15,15,15) | 1 | 1 | 2
  Red Blood Cells in Urine (n=5,7,6) | 1 | 0 | 0
  White Blood Cells in Urine (n=5,7,6) | 0 | 2 | 0

24. Secondary Outcome: Number of Participants With Out of Range Electrocardiogram (ECG) Intervals and Number of Participants With a Change From Baseline of Greater Than 30 Milliseconds in QT and QTcF
Description: Single 12-lead ECGs were obtained at screening, Day -1 of Period 1, and Days 4 and 7 of each treatment period after the participant had been supine for at least 5 minutes. Pulse Rate (PR), Complex of Q, R, S waves (QRS), and contraction of ventricle between the beginning of the Q wave and end of the T wave (QT) were measured in milliseconds (msec). QT was corrected by the Fridericia method (QTcF) and measured in msec. Baseline was Day -1 of first treatment period. Crossover study: same participant with out of range ECG intervals could be reported in multiple arms.
Time Frame: Day -1 first treatment period, Days 4 and 7 each treatment period
Population: Those participants who received any study medication and had available ECG data at baseline and Days 4 and 7 in each treatment period were analyzed.
Measure: Number; unit: participants
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Number analyzed (Participants) | 15 | 15 | 15
participants
  PR >200 msec (n=15,15,15) | 0 | 0 | 0
  QRS > 120 msec (n=15,15,15) | 0 | 0 | 0
  QT > 500 msec (n=15,15,15) | 0 | 0 | 0
  QTcF > 450 msec (n=15,15,15) | 0 | 0 | 0
  Change from Baseline >30 msec in QT (n=15,15,15) | 3 | 2 | 3
  Change from Baseline >30 msec in QTcF (n=15,15,15) | 0 | 0 | 0

25. Secondary Outcome: Mean Change From Baseline in Diastolic and Systolic Blood Pressure on Day 4 and Day 7
Description: Blood pressures were recorded at screening, Day -1 of Period 1, and Days 4 and 7 of each period. Blood pressure was measured after the participant had been seated quietly for at least 5 minutes and was measured in millimeters of mercury (mmHg). Baseline was last non-missing result with a collection date-time less than the date-time of the first active dose.
Time Frame: Screening, Day -1 first treatment period, Days 4 and 7 post treatment
Population: Those participants who received any study medication and had blood pressure data at baseline and post baseline were analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Number analyzed (Participants) | 15 | 15 | 15
mmHg
  Systolic BP Day 4 (n=15,15,15) | 0.9 (8.43) | -2.1 (10.67) | -2.9 (10.22)
  Systolic BP Day 7 (n=15,15,15) | 2.1 (8.03) | 3.7 (8.46) | 1.3 (8.87)
  Diastolic BP Day 4 (n=15,15,15) | -2.1 (6.64) | -3.3 (6.76) | -3.1 (5.70)
  Diastolic BP Day 7 (n=15,15,15) | -0.1 (8.34) | 0.0 (7.43) | -0.1 (6.58)

26. Secondary Outcome: Mean Change From Baseline in Heart Rate on Day 4 and Day 7
Description: Heart Rate was recorded at screening, Day -1 of Period 1, and Days 4 and 7 of each period. Heart Rate was measured after the participant had been seated quietly for at least 5 minutes and was measured in beats per minute (bpm). Baseline was last non-missing result with a collection date-time less than the date-time of the first active dose.
Time Frame: Screening, Day -1 first treatment period, Days 4 and 7 post treatment
Population: Those participants who received any study medication and had heart rate data at baseline and post baseline were analyzed.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Number analyzed (Participants) | 15 | 15 | 15
bpm
  Heart Rate Day 4 (n=15,15,15) | -4.3 (12.10) | -4.9 (11.46) | -5.5 (9.91)
  Heart Rate Day 7 (n=15,15,15) | -1.8 (10.09) | 0.4 (10.73) | -2.1 (10.17)

27. Secondary Outcome: Mean Change From Baseline in Respiration Rate on Day 4 and Day 7
Description: Respiration Rate was recorded at screening, Day -1 of Period 1, and Days 4 and 7 of each period. Respiration Rate was measured after the participant had been seated quietly for at least 5 minutes and was measured in respirations (breaths) per minute. Baseline was last non-missing result with a collection date-time less than the date-time of the first active dose.
Time Frame: Screening, Day -1 first treatment period, Days 4 and 7 post treatment
Population: Those participants who received any study medication and had respiration rate data at baseline and post baseline were analyzed.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Number analyzed (Participants) | 15 | 15 | 15
breaths per minute
  Respirate Rate Day 4 (n=15,15,15) | -0.7 (2.58) | -1.3 (1.87) | -1.4 (2.41)
  Respirate Rate Day 7 (n=15,15,15) | -0.4 (2.20) | -0.3 (2.41) | -0.5 (2.90)

28. Secondary Outcome: Mean Change From Baseline Temperature on Day 4 and Day 7
Description: Temperature was recorded at screening, Day -1 of Period 1, and Days 4 and 7 of each period and was measured in degrees centigrade (C). Baseline was last non-missing result with a collection date-time less than the date-time of the first active dose.
Time Frame: Screening, Day -1 first treatment period, Days 4 and 7 post treatment
Population: Those participants who received any study medication and had temperature data at baseline and post baseline were analyzed.
Measure: Mean (Standard Deviation); unit: C
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Number analyzed (Participants) | 15 | 15 | 15
C
  Temperature Day 4 (n=15,15,15) | -0.15 (0.432) | -0.14 (0.350) | -0.22 (0.399)
  Temperature Day 7 (n=15,15,15) | -0.20 (0.321) | -0.08 (0.328) | -0.17 (0.418)

ADVERSE EVENTS:
Time Frame: Day 1 to 30 days post last dose.
Description: Study initiated February 2014 and completed April 2014
Arm/Group | Treatment A: Apixaban + Placebo | Treatment B: Apixaban + Cofact (4-Factor PCC) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC)
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 5/15 | 2/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: Apixaban + Placebo (N=15) | Treatment B: Apixaban + Cofact (4-Factor PCC) (N=15) | Treatment C: Apixaban + Beriplex P/N (4-Factor PCC) (N=15)
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Traumatic Hematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Nightmare (Psychiatric disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.